CLINICAL TRIAL: NCT04856995
Title: Comparison of The Effects of Surgical Smoke on The Air Quality And on The Physical Symptoms of Operating Room Staff
Brief Title: Effect of Surgical Smoke on Air Quality
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: AIBU-SBF-GES-02
Record Dates: First submitted 2021-03-19; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Air Quality; Volatile Organic Compounds; Occupational Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- working in the operating: operating room workers exposed to surgical smoke
  Interventions: Other: exposure to surgical smoke during surgery
- working in internal units: Internal unit workers not exposed to surgical smoke

INTERVENTIONS:
Other: exposure to surgical smoke during surgery — No intervention was made. During the surgery, complaints and throat cultures were taken before and after exposure to surgical smoke. Simultaneously, 45 air samples are taken in the operating room before, during and after the operation.
  Groups: working in the operating

SUMMARY:
This study; It was planned to (1) determine the effect of surgical smoke on indoor air quality and (2) examine its effect on physical symptoms and throat culture results in operating room employees and compare it with those working in internal units.

DETAILED DESCRIPTION:
Background:This study is a experimental study. The aim of this study is; to determine the effect of surgical smoke containing toxic chemicals on indoor air quality and to examine the physical symptoms of employees in the operating room.

Method:It was carried out in general surgery operating room between June 2020 and July 2020 In the study, 45 air samples were taken from the with active sampling method before, during and after surgery. Physical complaints of 19 people working in the operating room were asked and throat cultures were taken before and after surgery. These results were compared with those working in internal units. Data were analyzed using a statistics program.

ELIGIBILITY:
Inclusion Criteria:

* Health workers in operating room

Exclusion Criteria:

* those with chronic diseases such as Chronic Obstructive Pulmonary Disease, Asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health workers in hospital
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
AIR UALITY IN OPERATING ROOM | 29/06/2020- 20/07/2020
  Surgical smoke contains cellular materials including polycyclic aromatic hydrocarbons (PAH) and volatile organic compounds (VOC) from carcinogenic chemicals.In the study, 45 air samples were taken from the general surgery operating room with active sampling method before, during and after surgery
THE PHYSICAL SYMPTOMS | 29/06/2020- 20/07/2020
  Physical complaints of 19 people working in the general surgery operating room were asked and throat cultures were taken before and after surgery. These results were compared with those working in internal units.

CONTACTS AND LOCATIONS:
Overall Officials: GANİME E SOYSAL, Study Director — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal Üniversitesi/Sağlık Bilimleri Fakültesi, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
STUDY PROTOCOL Data collection process
  Determining the effect of surgical smoke on air quality Taking air samples in the general surgery operating room (n: 45)
  1. Example: 45 minutes before the start of the operation
  2. Example: 45 minutes from the beginning of the skin incision
  3. Example: 45 minutes after the operations are over
  Determination of Physical Symptoms Caused by Surgical Smoke on Employees and Comparison
  Physicians and nurses in internal units control group(n: 20)
  Information Form Throat culture
  Case group (n: 19) Physicians and nurses exposed to surgical smoke in the general surgery operating room
  1. Before starting the operation Information form Throat culture
  2. After the surgery is over Information Form Throat culture
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When article is published in the journal
Access Criteria: Article is published in the journal

REFERENCES:
- [Background] Ulmer BC. The hazards of surgical smoke. AORN J. 2008 Apr;87(4):721-34; quiz 735-8. doi: 10.1016/j.aorn.2007.10.012. PMID 18461735
- [Background] Okoshi K, Kobayashi K, Kinoshita K, Tomizawa Y, Hasegawa S, Sakai Y. Health risks associated with exposure to surgical smoke for surgeons and operation room personnel. Surg Today. 2015 Aug;45(8):957-65. doi: 10.1007/s00595-014-1085-z. Epub 2014 Nov 25. PMID 25421864
- [Background] Choi SH, Kwon TG, Chung SK, Kim TH. Surgical smoke may be a biohazard to surgeons performing laparoscopic surgery. Surg Endosc. 2014 Aug;28(8):2374-80. doi: 10.1007/s00464-014-3472-3. Epub 2014 Feb 26. PMID 24570016
- [Background] Tramontini CC, Galvao CM, Claudio CV, Ribeiro RP, Martins JT. [Composition of the electrocautery smoke: integrative literature review]. Rev Esc Enferm USP. 2016 Feb;50(1):148-57. doi: 10.1590/S0080-623420160000100019. Portuguese. PMID 27007432
- [Background] Ilce A, Yuzden GE, Yavuz van Giersbergen M. The examination of problems experienced by nurses and doctors associated with exposure to surgical smoke and the necessary precautions. J Clin Nurs. 2017 Jun;26(11-12):1555-1561. doi: 10.1111/jocn.13455. Epub 2017 Mar 20. PMID 27345749

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04856995/Prot_SAP_ICF_000.pdf